CLINICAL TRIAL: NCT03196583
Title: Open Label Pilot Exploratory Study of a New Mandibular Oral Device for Mild to Moderate Obstructive Sleep Apnea: The BVL Project
Brief Title: Efficacy of a Novel MAD in OSA
Acronym: BVL Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mauro Manconi (Other)
Responsible Party: Sponsor-Investigator, Mauro Manconi, Head of Sleep and Epilepsy Center, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3184, BASEC 201700317
Record Dates: First submitted 2017-06-19; First posted 2017-06-23 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Sleep Apnea, Obstructive; Apnea, Obstructive; OSA; OSAH; Obstructive Sleep Apnea; Obstructive Sleep Apnea Syndrome
Keywords: obstructive sleep apnea syndrome; video-polysomnography; mandibular advancement device; oral device; cephalometry
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective, open-label, interventional, exploratory pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm study (Experimental): Velo-Lingual Bite (BVL)
  Interventions: Device: Velo-Lingual Bite (BVL)

INTERVENTIONS:
Device: Velo-Lingual Bite (BVL) — The administration of the device will proceed according to both the essential requirements of the European directives concerning medical devices (Annex I and X of directive 93/42/EEC) and the clinical practice standards and guidelines provided by the AASM and AASDM. These include the obtainment of alginate impression of both jaws and an interocclusal record, with the mandible at 50% of its maximal protrusive position. Since no single standard titration protocol is available, progressive mandibular advancement will be conducted according to the best available medical standard.

SUMMARY:
Oral appliances (OA) have emerged as an alternative to continuous positive airway pressure (CPAP) for obstructive sleep apnea (OSA) treatment. The most commonly used OA reduces upper airway collapse by advancing the mandible (mandibular advancement devices, MAD).

There is a strong evidence base demonstrating that MADs improve OSA in the majority of patients, including some with more severe disease. However, MADs are not efficacious for all, with approximately one-third of patients experiencing no therapeutic benefit. Patients often prefer MADs to gold-standard CPAP treatment. Head-to-head trials confirm CPAP is superior in reducing OSA parameters on polysomnography; however, this greater efficacy does not necessarily translate into better health outcomes in clinical practice. Comparable effectiveness of MADs and CPAP has been attributed to higher reported nightly use of MADs, suggesting that inferiority in reducing apnoeic events may be counteracted by greater treatment adherence.

The MAD in study, called Bite-Velo Linguale (BVL), features a novel monobloc device including a tongue retainer, a suction cavity that maintains the tongue down onto the mouth floor in order to prevent it from raising towards the hard palate, and therefore increasing the retro lingual aerial space. Its design requires the presence of only four occlusal points, allowing for a direct anchorage onto the mandibular bone, thus reducing the risk for occlusal changes, tooth loosening and the development of an anterior cross bite, which represent some of the major long-term adverse effects of oral appliances.

MADs are generally well tolerated, although short-term adverse effects during acclimatization are common. Long-term dental changes do occur, but these are for the most part subclinical and do not preclude continued use. The BVL in study features technological advances aimed at preventing long-term dental changes, as well as improving tolerability and easiness of use.

DETAILED DESCRIPTION:
The MAD in study features a novel monobloc device including a tongue retainer, a suction cavity to push the tongue down onto the mouth floor, thus preventing its lifting towards the hard palate, which improves retro lingual dimensions. Its design requires the presence of only four occlusal points, allowing for a direct anchorage onto the mandibular bone, thus reducing the risk for occlusal changes, tooth loosening and the development of an anterior cross bite, which represent the major long-term adverse effects of oral appliances.

MADs, as well as CPAP, represent the first choice treatment for mild-to-moderate OSAH. In several countries, as well as in Switzerland, health insurances cover the costs of MAD production in patients with mild-to-moderate OSAH or in severe OSAH patients who did not tolerate CPAP previously (as specified in the federal Mittel und Gegenständeliste (MiGeL), Position L 23.26.01.00.1).

Three main novelties justify the experimentation of this new MAD: a monobloc design, the combination with a tongue retainer and a potential future lower cost of production compared to the devices available on the market today.

The device will be designed, manufactured and used under the conditions and for the purposes intended. Thus, it will not compromise the clinical condition or the safety of patients, or the safety and health of users or, where applicable, other persons. Any risks, which may be associated with its intended use, constitute acceptable risks when weighed against the benefits to the patient and are compatible with a high level of protection of health and safety.

The administration of the device will proceed according to both the essential requirements of the European directives concerning medical devices (Annex I and X of directive 93/42/EEC) and the clinical practice standards and guidelines provided by the AASM and AASDM. These include the obtainment of alginate impression of both jaws and an interocclusal record, with the mandible at 50% of its maximal protrusive position. Since no single standard titration protocol is available, progressive mandibular advancement will be conducted according to the best available medical standard.

Monocentric, prospective, open-label, interventional, exploratory pilot study.

Patients aged 18-65 years who received a video-polysomnographic diagnosis of mild-to-moderate OSA (AHI between 5/h and 30/h) within three months will be screened and recruited at the Sleep and Epilepsy Center in Lugano. An ENT evaluation including a Müller maneuver and a calculation of the Mallampati Score must have been performed in order to rule out significant ENT comorbidities (See Section 7.1 Eligibility Criteria).

At Visit 1 (week 1: 7+3 days), performed by either Prof. Manconi or Dr. Chiaro, inclusion and exclusion criteria will be checked. Eligible patients will be included in the study.

Proof that a video-polysomnographic diagnosis of mild-to-moderate OSA was reached and that significant oropharyngeal disease was ruled out by means of fibro endoscopic evaluation, performed by a trained Ear, Nose & Throat (ENT) specialist in the last three months will be obtained.

During the visit, overall sleep quality and excessive daytime sleepiness will be evaluated by means of the Pittsburgh Sleep Quality Index (PSQI) and the Epworth Sleepiness Scale (ESS) (See Appendix 2).

At any time within Visit 1 and 2, (weeks 1 to 2, 14+3 days), the patient will undergo a head-CT scan. Patients will be scheduled for a CT scan of the oropharynx region at the Radiology Department of the Ospedale Civico of Lugano. CT scans (CT Siemens SOMATOM Definition Edge).will be performed in awake supine patients with their heads in a neutral position and will be repeated in the same session with and without the MAD. Subsequently, post-processing measurements of the upper airway will be calculated with a dedicated CT workstation.

At Visit 2 (week 2: 7+3 days), subjects will undergo odontological evaluation, performed by Dr Ciocco. This includes a first general clinical evaluation, the obtainment of alginate dental impressions (Blueprint creme, dust-free alginate impression material, manufactured by Dentsply® DeTrey GmbH 78467 Konstanz, Germany) with dental impression trays, the calculation of the dental facebow with an occlusal fork and of the bite with dental wax casts.

Weeks 3 to 4 (14+3 days) are the timeframe allotted to medical device production, which will be carried out by Mr Frigerio. Dental impressions will be modelled into chalk casts. Both casts will be then fixed on a dental articulator, so that different orthodontic measures can be calculated and the BVL will be produced out of resin (Palapress, powder+ liquid, Heraeus Kulzer GmbH, Grüner Weg 11, D-63450 Hanau) directly on the chalk casts, obtained from the patient's dental impression.

Once roughly finished, the two splints will be held together by means of an integrated advancement system composed by two stainless steel positioning holding screws (one left, one right) two serrated housing nuts (one left, one right), both produced by Leone SPA, Sesto Fiorentino, Italy, as well as two Dolder® system bars (one male, one female, two per side), produced by Cendres+Metaux SA, Biel/Bienne, Switzerland. This coupling system enables the horizontal (forwards) sliding of the lower splint on the upper splint, thus allowing mandibular advancement. The metal and resin parts are glued together with a primer produced by SHOFU Dental GmbH, Ratingen, Germany.

The BVL also features a tongue retainer, which will be completed by small holes on its anterior part in order to allow enhanced breathing and saliva excretion.

The BVL will then be finished, perfected and polished. A unique identification number and the BVL trademark will be printed on the BVL.

See Appendix 1 for technical and commercial details regarding used materials and their related available safety data.

At visit 3 (week 5-6: 7+3 days): the BVL will be then administered at 50% of mandibular advancement by Dr Ciocco, based on calculations of the patient's maximal mandibular protrusion. Immediate tolerability and side effects (i.e: myofacial pain, temporo-mandibular tension) will be checked by means of a semi-structured self-administered questionnaire (See Appendix 3) and duly noted.

If the patient experiences important side effects at this stage, he will discontinue the study.

At Visit 4 (week 7: 7+3 days), Dr Ciocco will perform further mandibular advancement to 60% of the calculated maximal mandibular protrusion by activating the integrated advancement system. Tolerability, side effects and compliance will be assessed by means of a semi-structured self-administered questionnaire (See Appendix 3) and duly noted.

At Visit 5 (week 8: 7+3 days), Dr Ciocco will perform further mandibular advancement to 70% of the calculated maximal mandibular protrusion by again activating the integrated advancement system. Tolerability, side effects and compliance will be assessed by means of a semi-structured self-administered questionnaire (See Appendix 3) and duly noted.

At Visit 6 (week 9 to 10, 14+3 days), the patient will undergo VPSG recording and a head-CT scan. Patients will be scheduled for a CT scan of the oropharynx region at the Radiology Department of the Ospedale Civico of Lugano. CT scans (CT Siemens SOMATOM Definition Edge).will be performed in awake supine patients with their heads in a neutral position and will be repeated in the same session with and without the MAD. Subsequently, post-processing measurements of the upper airway will be calculated with a dedicated CT workstation. At this point, tolerability, side effects and compliance will be assessed by means of a semi-structured self-administered questionnaire (See Appendix XXX) and duly noted.

If, at any point from MAD administration (Visit 3) to achievement of 70% mandibular protrusion (Visit 5), any serious side effect occurs, the patient will stop mandibular advancement and return to the previous level of mandibular protrusion, at which no side effects were experienced. He or she will then proceed directly to VPSG and Head-CT and then leave the study.

At the final evaluation (Visit 7, week 11), the patient will meet with the investigator again. PSQI and ESS will be administered to assess overall sleep quality and daytime sleepiness. Overall tolerability, side effects and compliance will be assessed by means of a semi-structured self-administered questionnaire (See Appendix 3) and duly noted. The custom-made MAD will be left with the patient free of charge.

We plan to include 20 study subjects. This study does not comply study groups, comparators or placebo. All subjects will receive treatment with MAD. For each patient, as described above, we plan a study duration of a maximum of 11 weeks. A shorter duration is foreseen for subjects who cannot reach a 70% mandibular advancement because of TMJ tension or for dropouts.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old
* VPSG within the last three months
* Diagnosis of mild-to-moderate OSAS (AHI 5-30/h)
* At least 4 teeth present in the lower and upper arch
* Ability to protrude the mandible for at least 6 mm
* Informed Consent

Exclusion Criteria:

* Significant ENT disease

  * Tonsillar hypertrophy
  * Uvulopalatopharyngoplasty (UPPP)
  * Palatoschisis
  * Neoplastic lesions
* Other neurological disorders

  * Trigeminal neuralgia
  * Myofacial pain dysfunction (MPD)
  * Central Sleep Apnea
  * Limited mental capacity
* Obesity (BMI > 30 kg/m2)
* Concomitant sleep-disordered breathing treatment (CPAP and/or positional therapy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Reduction in pathological breathing events | Weeks 9 to 10
  The primary outcome is the numerical reduction in pathological sleep-related breathing events because of treatment with the BVL, as measured by changes in the AHI.

SECONDARY OUTCOMES:
Treatment-Emergent Side effects | At weeks 5, 7, 8, 9, 11
  Subjectively by means of a semi-structured self-administered questionnaire covering the following aspects: Usage (nights/week; hours/night); Side effects/reasons for interrupting usage; Visual Analogue Scale for Pain (VAS Pain); Visual Analogue Scale for Satisfaction (VAS Satisfaction).
Usage (number of nights/week) | At weeks 5, 7, 8, 9, 11
  Subjectively by means of a semi-structured self-administered questionnaire covering the following aspects: Usage (nights/week; hours/night); Side effects/reasons for interrupting usage; Visual Analogue Scale for Pain (VAS Pain); Visual Analogue Scale for Satisfaction (VAS Satisfaction).
Usage (number of hours/night) | At weeks 5, 7, 8, 9, 11
  Subjectively by means of a semi-structured self-administered questionnaire covering the following aspects: Usage (nights/week; hours/night); Side effects/reasons for interrupting usage; Visual Analogue Scale for Pain (VAS Pain); Visual Analogue Scale for Satisfaction (VAS Satisfaction).
Pain | At weeks 5, 7, 8, 9, 11
  Subjectively by means of a semi-structured self-administered questionnaire covering the following aspects: Usage (nights/week; hours/night); Side effects/reasons for interrupting usage; Visual Analogue Scale for Pain (VAS Pain); Visual Analogue Scale for Satisfaction (VAS Satisfaction).
Satisfaction with the device | At weeks 5, 7, 8, 9, 11
  Subjectively by means of a semi-structured self-administered questionnaire covering the following aspects: Usage (nights/week; hours/night); Side effects/reasons for interrupting usage; Visual Analogue Scale for Pain (VAS Pain); Visual Analogue Scale for Satisfaction (VAS Satisfaction).
Modification in global AHI | Weeks 9 to 10
  Modification of the apnea-hypopnea index, measured as the objective numerical difference in the parameter between baseline PSG to final PSG
Modification in NREM AHI | Weeks 9 to 10
  Modification of non-REM-sleep apnea-hypopnea index, measured as the objective numerical difference in the parameter between baseline PSG to final PSG
Modification in REM AHI | Weeks 9 to 10
  Modification of REM-sleep apnea-hypopnea index, measured as the objective numerical difference in the parameter between baseline PSG to final PSG
Modification in supine AHI | Weeks 9 to 10
  Modification of the supine apnea-hypopnea index, measured as the objective numerical difference in the parameter between baseline PSG to final PSG
Modification in ODI≥3% | Weeks 9 to 10
  Modification of the oxygen desaturation index, measured as the objective numerical difference in the parameter between baseline PSG to final PSG
Modification in RDI | Weeks 9 to 10
  Modification of respiratory distress index, measured as the objective numerical difference in the parameter between baseline PSG to final PSG
Modification in T90 | Weeks 9 to 10
  Modification of the time spent at an oxygen saturation below 90%, measured as the objective numerical difference in the parameter between baseline PSG to final PSG
Modification in snoring time | Weeks 9 to 10
  Modification of the snoring time, measured as the objective numerical difference in the parameter between baseline PSG to final PSG
Modification in TST | Weeks 9 to 10
  Modification of the total sleep time, measured as the objective numerical difference in the parameter between baseline PSG to final PSG
Modification in SL | Weeks 9 to 10
  Modification of the sleep latency, measured as the objective numerical difference in the parameter between baseline PSG to final PSG
Modification in SE | Weeks 9 to 10
  Modification of the sleep efficiency, measured as the objective numerical difference in the parameter between baseline PSG to final PSG
Modification in WASO | Weeks 9 to 10
  Modification of the wake after sleep onset, measured as the objective numerical difference in the parameter between baseline PSG to final PSG

OTHER OUTCOMES:
Overall Sleep Quality | At week 1 and week 11
  Subjectively with the Pittsburgh Sleep Quality Index
Daytime Somnolence | At week 1 and week 11
  Subjectively with the Epworth Sleepiness Scale
Modification in upper airway volume | At week 1 and week 11
  The modification in upper airway volume induced by the MAD will be measured by cross-sectional CT imaging of the oropharynx region.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Manconi, MD, PhD, Principal Investigator — Sleep and Epilepsy Center, Neurocenter of Southern Switzerland, Ospedale Civico di Lugano, Ente Ospedaliero Cantonale
Locations (1):
- Sleep and Epilepsy Center, Neurocenter of Southern Switzerland, Ospedale Civico di Lugano, Ente Ospedaliero Cantonale, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to researchers not pertaining to this project.